CLINICAL TRIAL: NCT01907893
Title: Improving Activity and Quality of Life Following Orthopaedic Trauma: The Trauma Collaborative Care Study (TCCS)
Acronym: TCCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Major Extremity Trauma Research Consortium (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: METRC - TCCS
Record Dates: First submitted 2013-07-09; First posted 2013-07-25 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Severe Orthopedic Trauma
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trauma Collaborative Care Plus Treatment as Usual (Experimental): Three components: (1) Services provided through the Trauma Survivors Network (TSN) Program; (2) Provider training to reinforce referral to and use of TSN programs; and (3) Enhancement of collaborative care through the use of a TSN Coordinator (TSN-C).
  Interventions: Behavioral: Trauma Collaborative Care Plus Treatment as Usual
- Treatment as Usual (No Intervention): Study patients treated at Control Sites will have access to all services typically available to patients treated at these centers.

INTERVENTIONS:
Behavioral: Trauma Collaborative Care Plus Treatment as Usual
  Other Names: TSN
  Arms: Trauma Collaborative Care Plus Treatment as Usual

SUMMARY:
The study uses a multi-site, cluster design to determine the effectiveness of an intervention based on a Trauma Collaborative Care (TCC) model in improving patient outcomes for persons with severe orthopedic trauma and enhancing both patient and provider satisfaction with overall care. The study will also determine the cost and cost-effectiveness of the intervention.

Primary Hypothesis: Compared to standard treatment alone, access to the TCC Program plus standard treatment will result in lower rates of the composite outcome (i.e. positive for poor function, depression, and/or PTSD).

Secondary Hypotheses: Compared to standard treatment alone, access to the TCC Program plus standard treatment will result in lower levels of pain and higher rates of return to usual major activity and higher levels of health related quality of life. In addition, both primary and secondary outcomes will correlate strongly with the intermediate outcome of self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients treated surgically for one or more orthopaedic injuries with initial admission to the trauma service of the participating hospital
2. Ages 18-60 yrs inclusive
3. Length of Stay (LOS) >=5 days or >= 3 days with planned readmission for additional procedures
4. At least one orthopaedic injury of AIS 3 or greater (determination based on information available at the time of enrollment) resulting from a moderate to high energy force (e.g. motor vehicle or motorcycle crash, high fall). Injuries can include those to the upper or lower extremities, pelvis/acetabulum or spine.
5. Traumatic amputations of the upper or lower extremities (excluding amputations to fingers or toes)

Exclusion Criteria:

1. Initial admission to non-trauma service.
2. Peri-prosthetic fractures of the femur, regardless of etiology
3. Patient eligible for the METRC OUTLET Study, i.e. patient with:

   1. Gustilo type III distal tibia and/or foot or type III B or C ankle fractures with fracture pattern consistent with one of OTA codes: 43B1.3, 43B2-B3, 43C, 44B, 44C, 81B2-B3, 82B, and 82C;
   2. Open or closed industrial foot crush injuries;
   3. Open or closed foot blast injuries.
4. Patient requiring a Legally Authorized Representative (as defined by an inability to answer the "Evaluation of Give Consent" questions)
5. Patient non-ambulatory due to an associated spinal cord injury
6. Patient non-ambulatory pre-injury
7. Non-English speaking
8. Patient diagnosed with a severe psychosis
9. Patient lives outside the hospital's catchment area and/or follow-up is planned at another medical center
10. Severe problems with maintaining follow-up expected (e.g. patients who are prisoners or homeless at the time of injury or those who are severely intellectually challenged).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 900 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Composite Outcome: A binary composite outcome comprised of patient reported assessments of function, depression and post traumatic stress (PTSD). | 12 months
  * Functional Status: the Short Musculoskeletal Functional Assessment (SMFA)
  * Depressive Symptoms : the nine item depression scale of the Patient Health Questionnaire (PHQ-9)
  * Post-Traumatic Stress: the PTSD Checklist, civilian version (PCL)

SECONDARY OUTCOMES:
Health Related Quality of Life | 6 weeks, 6 and 12 months
  • Veterans RAND 12 Item Health Survey (VR-12) and its utility based derivative, the VR-6D The 6 week assessment collects pre-injury Health related Quality of life
Return to Usual Activity | 6 weeks; 6 and 12 months
  Standard questions assessing usual major activity The 6 week assessment collects pre injury usual activity
Self Efficacy | Baseline; 6 weeks; 6 and 12 months
  Modified Self-Efficacy Scale
• Use and Satisfaction with TCC Program and its component services (TSN Questions) | 6 and 12 months
  for intervention group only
• Satisfaction with Overall Care | 6 and 12 months
  Short Form Patient Satisfaction Questionnaire (PSQ-18)
Patient productivity in work | 6 and 12 months
  • Work Productivity and Activity Impairment Questionnaire (WPAI)
Referral to TSN activities | 6 and 12 months
  A secondary provider reported outcome(assessed by review of Recovery Plan)
Provider satisfaction | 6 and 12 months
  • Provider satisfaction with care received by their patients in the inpatient and outpatient setting
Provider confidence | 12 months
  • Confidence in managing psychosocial factors related to orthopaedic trauma
Self reported service use | 6 and 12 months
  • Self-reported utilization data on number of inpatient visits, emergency department visits, and unscheduled outpatient surgeries related to study injuries
Intervention program costs | 12 months
  • Costs of the intervention based on costs to implement and sustain program

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Denver Health and Hospital Authority, Denver, Colorado
  - St Josephs Hospital, Tampa, Florida
  - Tampa General Hospital, Tampa, Florida
  - Methodist Hospital, Indianapolis, Indiana
  - University of Maryland/ R Cowley Adams Shock Trauma Center, Baltimore, Maryland
  - Spectrum Health/Orthopaedic Institutes of Michigan, Grand Rapids, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest Baprtist Medicla Center, Winston-Salem, North Carolina
  - Metro Health, Cleveland, Ohio
  - Vanderbilt Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center - HOUSTON, Houston, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia